CLINICAL TRIAL: NCT06824298
Title: Effect of TENS on Bladder Tenesmus-related Pain and Patient Comfort in the Early Postoperative Period After Urinary Surgery
Brief Title: Effect of TENS on Bladder Tenesmus-related Pain and Patient Comfort After Urinary Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Dr. Özlem İbrahimoğlu, Associate Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IstanbulMU8
Record Dates: First submitted 2025-02-02; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Urinary Surgery; Pain, Postoperative; Comfort
Keywords: Bladder tenesmus; Pain; Comfort; Nursing care
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Patients who were hospitalized for urinary surgery and met the sample selection criteria will be included in the experimental and control groups by block randomization method using the random numbers table on the computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS application group (Experimental): Before surgery: The socio-demographic data of the patients will be recorded. During surgery: After patients are taken to the operating room and anesthesia is induced, TENS electrodes will be attached to the paravertebral muscles at the level of Lumbar vertebrae 2, 3 and Sacral Vertebrae 2, 3. After the surgery is completed, TENS will be activated before the patient is woken up.
  TENS settings: In modulation type, medium intensity contractions will be given at a frequency ranging from 60-80 Hertz to 1-5 Hertz, with a current rate ranging from 50-100 microseconds to 150-200 microseconds.
  After surgery: TENS will continue to be applied to patients in the recovery room for 30 minutes after the surgery. Patients will be evaluated by researchers in terms of pain and comfort associated with bladder tenesmus at 0, 15 and 30 minutes in the recovery room and at 6, 12 and 24 hours in the postoperative ward.
  Interventions: Other: TENS
- Control group (No Intervention): Patients in the control group will receive standard care that includes all medical and non-medical treatments in the hospital. Nursing care, which is routinely applied to patients in the postoperative period, both in the recovery room and in the service, will be continued within the standard care. The patients will be evaluated by the researchers in terms of pain and comfort associated with bladder tenesmus at 0, 15 and 30 minutes in the recovery room and at 6, 12 and 24 hours in the postoperative ward.

INTERVENTIONS:
Other: TENS — Before surgery: The socio-demographic data of the patients will be recorded. During surgery: After patients are taken to the operating room and anesthesia is induced, TENS electrodes will be attached to the paravertebral muscles at the level of Lumbar vertebrae 2, 3 and Sacral Vertebrae 2, 3. After the surgery is completed, TENS will be activated before the patient is woken up.
  TENS settings: In modulation type, medium intensity contractions will be given at a frequency ranging from 60-80 Hertz to 1-5 Hertz, with a current rate ranging from 50-100 microseconds to 150-200 microseconds.
  After surgery: TENS will continue to be applied to patients in the recovery room for 30 minutes after the surgery. Patients will be evaluated by researchers in terms of pain and comfort associated with bladder tenesmus at 0, 15 and 30 minutes in the recovery room and at 6, 12 and 24 hours in the postoperative ward.
  Arms: TENS application group

SUMMARY:
Bladder tenesmu is defined as the need to urinate despite the person urinating and is associated with various causes such as bladder spasm, infection, stones, catheters. Catheters used in urinary surgeries can cause various complications, especially pain and discomfort. There is no sufficient study in the literature on bladder tenesmus caused by mechanical interactions related to urinary catheters, and this situation negatively affects patient comfort. Transcutaneous Electrical Nerve Stimulation (TENS) is an effective method of reducing pain with low-voltage electrical current. However, there are no studies on the application of TENS in the management of symptoms associated with bladder tenesmus after urinary surgery. This study aims to investigate the effect of TENS application on bladder tenesmus-related pain and patient comfort in the early postoperative period after urinary surgery.

DETAILED DESCRIPTION:
Bladder tenesmus is defined as the condition where a person still feels the need to urinate even though they have urinated. It may be caused by a tumor growing in the bladder or pelvis, or it may be associated with other bladder problems such as bladder spasm and discomfort, retention, infection, stones, clots, and catheters. During urological surgery, urinary catheters are placed in patients to ensure patency of the urinary tract, and these catheters usually remain in place until the patient is mobilized after surgery. Although urinary catheter-related problems are reported in the literature as short-term and long-term problems depending on the duration of the catheter, these problems are classified as infectious and non-infectious complications. The most common urinary catheter complications have been reported to include anaphylaxis, cytotoxicity and hypersensitivity, symptomatic bacterial infection, catheter obstruction, hematuria, mechanical trauma (perforation and urine leakage), urethral fistula and urethral stenosis. In a systematic review by Hollingsworth et al., where the results of 37 studies were evaluated, it was reported that non-infectious complications related to urinary catheters were much higher than infection-related complications. In a multicenter study by Saint et al., it was reported that infections constituted 10.5% of urinary catheter-related complications, while non-infectious complications constituted 55.4%, and these complications included pain and discomfort, hematuria, and urgent need to urinate. There are many studies on the successful application of non-pharmacological agents in pain treatment. One of these methods is Transcutaneous Electrical Nerve Stimulation (TENS). TENS is a method of applying controlled, low-voltage electrical current to the nervous system through electrodes placed on the skin and is widely used for postoperative pain control. Bladder tenesmus caused by a urinary catheter creates a feeling of a full bladder, causing pain and discomfort with symptoms of urgency and inability to urinate. This negatively affects the patient's comfort. Although urinary catheter-related complications have been extensively investigated, no comprehensive review has been conducted focusing on identifying and analyzing the complication of bladder tenesmia and urgency caused by mechanical interaction due to the physical contact of the urinary catheter. There is also no application in the literature to relieve symptoms associated with bladder tenesmus caused by Foley catheters in patients after urinary surgery. Therefore, this study was planned to investigate the effect of TENS application on pain and patient comfort associated with bladder tenesmus in the early postoperative period after urinary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* To undergo endoscopic urological surgery (Transurethral prostate resection/bladder surgery)
* Having an ASA score of 1-2
* Inserting a urinary catheter during surgery
* To be willing to participate in the study

Exclusion Criteria:

* To undergo emergency surgery
* Being under the age of 18
* Having an ASA score of 3 and above
* Having a urinary catheter inserted before surgery
* Not agreeing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
TENS | First 24 hours after surgery
  Change in pain score related to bladder tenesmus as measured by Visual Analog Scale (VAS) at 0, 15, and 30 minutes, and 6, 12, and 24 hours post-intervention.
TENS | First 24 hours after surgery
  Change in patient comfort score related to bladder tenesmus as measured by Numeric Rating Scale (NRS) at 0, 15, and 30 minutes, and 6, 12, and 24 hours post-intervention.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finegan, W. C., McGurk, A., O'Donnell, W., Pederson, J., & Rogerson, E. (2018). Tenezm. In Care of the Cancer Patient (pp. 196-197). CRC Press.
- [Background] Dellimore KH, Helyer AR, Franklin SE. A scoping review of important urinary catheter induced complications. J Mater Sci Mater Med. 2013 Aug;24(8):1825-35. doi: 10.1007/s10856-013-4953-y. Epub 2013 May 10. PMID 23661258
- [Background] Hollingsworth JM, Rogers MA, Krein SL, Hickner A, Kuhn L, Cheng A, Chang R, Saint S. Determining the noninfectious complications of indwelling urethral catheters: a systematic review and meta-analysis. Ann Intern Med. 2013 Sep 17;159(6):401-10. doi: 10.7326/0003-4819-159-6-201309170-00006. PMID 24042368
- [Background] Saint S, Trautner BW, Fowler KE, Colozzi J, Ratz D, Lescinskas E, Hollingsworth JM, Krein SL. A Multicenter Study of Patient-Reported Infectious and Noninfectious Complications Associated With Indwelling Urethral Catheters. JAMA Intern Med. 2018 Aug 1;178(8):1078-1085. doi: 10.1001/jamainternmed.2018.2417. PMID 29971436
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Bulut H, Erden S, Demir SG, Cakar B, Erdogan Z, Demir N, Ay A, Aydin E. The Effect of Cold Vapor Applied for Sore Throat in the Early Postoperative Period. J Perianesth Nurs. 2016 Aug;31(4):291-7. doi: 10.1016/j.jopan.2014.10.005. Epub 2016 Feb 24. PMID 27444760
- [Background] Erden, S., & Şenol Çelik, S. (2015). Bir elektro analjezi yöntemi: transkütan elektriksel sınır stimülasyonu ve hemşirenin rolleri. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi, 2(1), 50-60.
- [Background] Johnson, M. I. (2017). Pain Management and Clinical Effectiveness of TENS. Critical Reviews™ in Physical and Rehabilitation Medicine, 29(1-4).
- [Background] Vance CGT, Dailey DL, Chimenti RL, Van Gorp BJ, Crofford LJ, Sluka KA. Using TENS for Pain Control: Update on the State of the Evidence. Medicina (Kaunas). 2022 Sep 22;58(10):1332. doi: 10.3390/medicina58101332. PMID 36295493
- [Background] Song B, Chang Y, Li Y, Zhu J. Effects of Transcutaneous Electrical Acupoint Stimulation on the Postoperative Sleep Quality and Pain of Patients After Video-Assisted Thoracoscopic Surgery: A Prospective, Randomized Controlled Trial. Nat Sci Sleep. 2020 Oct 27;12:809-819. doi: 10.2147/NSS.S270739. eCollection 2020. PMID 33154688